CLINICAL TRIAL: NCT05903729
Title: Effects of Task Oriented Activities Based on Neurodevelopmental Therapy Principles on Trunk Control and Upper Extremity Function in Children With Spastic Diplegic Cerebral Palsy
Brief Title: Task Oriented Activities Based on NDT Therapy Principles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0711
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Cerebral Palsy
Keywords: CP, NDT therapy, task-oriented training, trunk control
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: It is a randomized control trial, used to compare conventional physiotherapt and neurodevelopmental therapy approaches on trunk control and upper extremity function in spastic diplegic cerebral palsy patients. subjects with spastic diplegic cerebral palsy meeting the predetermined inclusion and exclusion criteria will be divided into two groups using simple random sampling technique.
Who Masked: Participant
Masking Description: participants will get separate treatment protocols and possible efforts will be put to mask the both groups about their treatmaent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- neurodevelopmental therapy group (Experimental): in this group patients wil be treated with task oriented activities using neurodevelopmental therapy principles. This group will receive therapy session for 1 hour 6 days a week and for 8 weeks. total sessions will be 48. this group will receive task oriented neurodevelopmental therapy for 30 mins and next 30 mins it will receive conventional treatment.
  Interventions: Other: Neurodevelopmental therapy treatment
- conventional physiotherapy group (Experimental): in this group patients will be treated with conventional physiotherpy treatment protocol. this group will receive therapy session for one hour, 6 times in a week for 8 weeks. total therapy sessions will be 48. this group will receive 30 mins conventional physiotherapy treatment and 30 mins task oriented neurodevelopmental therapy.
  Interventions: Other: conventional physiotherapy

INTERVENTIONS:
Other: Neurodevelopmental therapy treatment — The group will receive NDT therapy
  Arms: neurodevelopmental therapy group
Other: conventional physiotherapy — conventional physiotherapy
  Arms: conventional physiotherapy group

SUMMARY:
Cerebral palsy (CP) is one of the primary causes of disability effecting majority of pediatric population. Cerebral Palsy is considered a neurological disorder caused by a non-progressive brain injury or malformation that occurs while the child's brain is under development. The worldwide incidence of cerebral palsy is it affects three to four individuals out of 1000 individuals in the general population. Cerebral palsy has different types depending upon the severity of disease or the area of the body it is affecting. Amongst the different types of CP, spastic diplegia is the most common type which mainly affects the lower extremities and lesser extent to upper extremities. It mainly affects functional performance and gait.

DETAILED DESCRIPTION:
This study will be conducted on 20 subjects which would be equally divided into experimental and control groups. Trunk control measurement scale (TCMS) and quality of upper extremity skills test (QUEST) will be the tools used in this study. Pre and post values of the effects of intervention will be evaluated. The significance of this study is that it will help us how to improve trunk control and upper extremity function in spastic dipegic children. Data will be analyzed using SPSS 22.0. Mean and standard deviation will be calculated. Appropriate statistical test will be used after checking normality of data.

ELIGIBILITY:
Inclusion Criteria:

* • Children with spastic diplegic cerebral palsy with age between 6 to 12 years.

  * Children with spastic diplegic cerebral palsy who are able to follow verbal commands.
  * Children with spastic diplegic cerebral palsy having level II or III of gross motor function classification system.

Exclusion Criteria:

* • Children who are uncooperative and having neurological deficit.

  * Children with hearing deficit.
  * Children with epilepsy.
  * Children with cardiac anomalies which effect exercise tolerance.
  * Children having less than 6-month post-orthopedic surgery.
  * Children having less than 6-month post-botulinum toxin injection (BOTOX).

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
The trunk control measurement scale | 8 weeks
  The Trunk Control Measurement Scale is a clinical tool to measure trunk control in children with cerebral palsy.

SECONDARY OUTCOMES:
The Quality of Upper Extremity Skills Test (QUEST) | 8 weeks
  The Quality of Upper Extremity Skills Test is an outcome measure designed to evaluate movement patterns and hand function in children with cerebral palsy.

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha tul Fatima, MS, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sah AK, Balaji GK, Agrahara S. Effects of Task-oriented Activities Based on Neurodevelopmental Therapy Principles on Trunk Control, Balance, and Gross Motor Function in Children with Spastic Diplegic Cerebral Palsy: A Single-blinded Randomized Clinical Trial. J Pediatr Neurosci. 2019 Jul-Sep;14(3):120-126. doi: 10.4103/jpn.JPN_35_19. Epub 2019 Sep 27. PMID 31649770
- [Background] Talgeri AJ, Nayak A, Karnad SD, Jain P, Tedla JS, Reddy RS, Sangadala DR. Effect of Trunk Targeted Interventions on Functional Outcomes in Children with Cerebral Palsy- A Systematic Review. Dev Neurorehabil. 2023 Apr;26(3):193-205. doi: 10.1080/17518423.2023.2193265. Epub 2023 Apr 5. PMID 37021364